CLINICAL TRIAL: NCT01334047
Title: Phase I/II Trial of Vaccine Therapy in Recurrent Platinum Sensitive Epithelial Ovarian Cancer Patients Using Autologous Dendritic Cells Loaded With Amplified Ovarian Cancer Stem Cell mRNA, hTERT and Survivin.
Brief Title: Trial of Vaccine Therapy in Recurrent Platinum Sensitive Ovarian Cancer Patients
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study needed to be terminated due to new knowledge about cancer vaccines. A new protocol with an expected more efficient vaccine is currently being written.
Sponsor: Steinar Aamdal (Other)
Responsible Party: Sponsor-Investigator, Steinar Aamdal, MD, PhD, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DC-006
Record Dates: First submitted 2011-03-30; First posted 2011-04-12 (Estimated); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Recurrent Epithelial Ovarian Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- DC vaccine (Experimental): Dendritic cells loaded with amplified ovarian cancer stem cell mRNA, hTERT and Survivin.
  Interventions: Biological: DC-006 vaccine

INTERVENTIONS:
Biological: DC-006 vaccine — Vaccine is administered every 4 weeks during the first year. Only patients that show immunological response will continue vaccination every months during the 2nd and 3rd year.
  Other Names: Dendritic cell vaccine

SUMMARY:
In this study the investigators will include patients with relapsed epithelial ovarian cancer. In spite of increased rates of complete response to initial chemotherapy, most patients with advanced ovarian cancer relapse and succumb to progressive disease. Immunotherapy may have potential for consolidation therapy. Dendritic cell vaccine is well toleranted in previous studies, with minor side effects and no serious adverse events registrated In this study, patients will receive DC-vaccine therapy after response to platinum treatment at relapse. The investigtors include patients in good clinical condition with no severe symptoms of the disease. If patients relapse during vaccine treatment, they will be discontinued from the study.

The investigators have included hTERT- and survivin mRNA in addition to amplified cancer stem cell mRNA in the vaccine.

DETAILED DESCRIPTION:
Study Period:

* Estimated date of first patient enrolled: First quarter of 2011
* Anticipated recruitment period: 3 years
* Estimated date of last patient completed: First quarter of 2017, follow up to 2022.

Treatment duration:

Patients will receive intradermal immunization once a week for 4 weeks followed by monthly "vaccine boost" during the first year. Patients that show immunological response will continue with vaccination every month the second and third year or as long as there is vaccine available. The patients will have follow up for 5 years or until progression of disease as evaluated by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed epithelial ovarian cancer. Histologic documentation of the original primary tumor is required via pathology report.
* Completed first line treatment (surgery and adjuvant or neoadjuvant treatment with carboplatine and paclitaxel)
* Relapsed and platinum sensitive epithelial ovarian carcinoma patients with response to chemotherapy in recurrent disease
* If surgery is indicated, the patient should be surgically treated and then starts vaccination with a minimum interval of 28 days.
* Must be ambulatory with an ECOG performance status 0 or 1.
* Life expectancy ≥ 6 months
* Must be of 18-75 years of age
* Must have lab values as the following:

  * ANC ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Hb ≥ 9 g/dL (≥ 5.6 mmol/L)
  * Creatinine ≤ 140 μmol/L (1.6 mg/dL); if borderline, the creatinine clearance ≥ 40 mL/min
  * Bilirubin within the upper limit of normal
  * ASAT and ALAT ≤ 2.5 the upper limit of normal
  * Albumin levels above lower normal value
* If the patient has preserved fertility after primary treatment, she must practice adequate contraception during the study treatment
* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Eligible to otherwise curative treatment.
* History of prior malignancy, other than ovarian cancer, within the last 5 years, with the exception of curatively treated basal cell carcinoma and cancer in situ cervix uteri.
* Prior surgery within the past 28 days
* Clinical ascites or metastatic pleural fluid
* Active infection requiring antibiotic therapy.
* Have known active central nervous system (CNS) or leptomeningeal metastasis (brain metastasis). Patients with signs or symptoms of neurological compromise should have appropriate radiographic imaging performed before study entry to rule out brain metastasis.
* Significant cardiac or other medical or mental illness that would limit activity or survival, such as severe congestive heart failure, unstable angina, serious cardiac arrhythmia or psychosis.
* Pregnancy or lactation
* Previous adverse reactions to vaccines such as asthma, anaphylaxis or other serious reactions.
* History of immunodeficiency or autoimmune disease such as but not limited to rheumatoid arthritis, systemic lupus erythematosus, scleroderma, polymyositis-dermatomyositis, juvenile onset insulin dependent diabetes, or a vasculitic syndrome.
* Positive for syphilis (treponema pallidum), HIV, Hepatitis B and C tests
* Use of systemic glucocorticoids.
* Prior anti-cancer treatment, including radiotherapy, chemotherapy immunotherapy and/or immunomodulating agents stopped for less than 4 weeks before first study treatment administration. Anti hormonal treatment, such as Tamoxifen, may continue until first study treatment administration.
* Any reason why, in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-04; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of adverse events | Up to 3 years
  Patients are coming every 4 weeks to the site during the 3 years vaccination period and every 6 months during the 5 years follow up period.
  Biochemistry and hematology results, vital signs and ECOG performance status will be measured at those timepoints during vaccination period.

SECONDARY OUTCOMES:
Determine immunological response to the vaccine (induction of specific T-cell response) | 8, 12 weeks after start of vaccination and every 3 months thereafter
Determine time of disease progression and survival time. | Every 4 weeks during vaccination and every 3-6 months during follow up
  Clinical response will be evaluated via:
  * measurement of CA-125 every 4 weeks
  * physical examination every 3rd months during vaccination
  * CT taken every 3rd months during vaccinaton and every 3-6 months during follow up.
Treatment free interval | up to 5 years after vaccination
  Start date of new antineoplastic therapy since discontinuation of the study will be recorded to capture information regarding treatment free interval.

CONTACTS AND LOCATIONS:
Overall Officials: Steinar Aamdal, M.D PhD Prof, Principal Investigator — Oslo University Hospital - Norwegian Radium Hospital
Locations (1):
- Oslo University Hospital- Norwegian Radium Hospital, Oslo, Norway